CLINICAL TRIAL: NCT00367198
Title: Protein Supplementation in Dialysis Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of enrollment
Sponsor: Vanderbilt University (Other)
Responsible Party: Alp Ikizler, MD, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 060587
Record Dates: First submitted 2006-08-18; First posted 2006-08-22 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2011-07

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): 30 ml per serving
  Interventions: Dietary Supplement: Pro-Stat
- 2 (Active Comparator): 60 ml per serving
  Interventions: Dietary Supplement: Pro-Stat
- 3 (No Intervention): chronic hemodialysis patients
- 4 (No Intervention): healthy subjects

INTERVENTIONS:
Dietary Supplement: Pro-Stat — two separate oral ingestions of nutrition supplement (either 30 ml per serving or at 60 ml per serving) during the hemodialysis session
  Arms: 1; 2

SUMMARY:
The mortality rate in chronic hemodialysis (CHD) patients remains excessively high and approaches 21% per year. Among the many factors that adversely affects patient outcome is uremic malnutrition, a unique form of deranged nutritional status. It is associated with increased hospitalization and death risk in CHD patients. Several measures have been identified to prevent uremic malnutrition in CHD patients, including efforts to optimize dialysis regimen and dietary protein and energy intake. A large number of CHD patients suffer from uremic malnutrition in spite of these aggressive measures. The inevitable protein catabolic effects of the hemodialysis procedure are important factors leading to increased prevalence of uremic malnutrition. Preliminary data suggest that oral nutritional supplementation administered during the hemodialysis procedure counteracts these protein catabolic effects and leads to net protein anabolism in the acute setting. In this proposal, we hypothesize that Pro-Stat, a high nitrogen, enzyme-hydrolyzed, tryptophan-fortified, collagen protein supplement will reverse the net protein catabolism observed during hemodialysis procedure.

ELIGIBILITY:
Inclusion criteria:

* On hemodialysis for more than 3 months, on a thrice weekly hemodialysis program.
* Adequately dialyzed (Kt/V > 1.2).
* Age 18-75

Exclusion criteria:

* Pregnant women.
* Severe unstable underlying disease besides commonly associated with end stage renal disease. Cardiac patients that are stable will be included.
* Patients hospitalized within the last month prior to the study.
* Patients with malfunctioning arterial-venous access [recirculation and/or blood flow < 500 ml/min for an arterial-venous graft (AVG) or <400 ml/min for an arterial-venous fistula (AVF)] Patients receiving steroids and/or other immunosuppressive agents.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2006-08; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
net muscle protein balance | 10 hours

CONTACTS AND LOCATIONS:
Overall Officials: Alp Ikizler, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Mah JY, Choy SW, Roberts MA, Desai AM, Corken M, Gwini SM, McMahon LP. Oral protein-based supplements versus placebo or no treatment for people with chronic kidney disease requiring dialysis. Cochrane Database Syst Rev. 2020 May 11;5(5):CD012616. doi: 10.1002/14651858.CD012616.pub2. PMID 32390133